CLINICAL TRIAL: NCT03088098
Title: Randomized Comparison of Left Atrial Appendage Occlusion vs Standard Medical Therapy in Patients in Atrial Fibrillation Undergoing Transfemoral Transcatheter Aortic Valve Implantation: The TAVI LAAO Trial
Brief Title: Comparison of Left Atrial Appendage Occlusion vs Standard Medical Therapy in Patients in AF Undergoing TAVI
Acronym: TAVI/LAAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0459
Record Dates: First submitted 2016-11-22; First posted 2017-03-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Aortic Stenosis
Keywords: left atrial appendage occlusion; transcatheter aortic valve implantation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): Patient receiving LAAO
  Interventions: Device: LAAO
- Control (No Intervention): Patient undergoing medical therapy for stroke prevention

INTERVENTIONS:
Device: LAAO — Left atrial appendage occlusion for stroke prevention
  Arms: Treatment

SUMMARY:
Study category and Rationale Clinical study, Category A.

Clinical Phase: Post market study

Background and Rationale: Left atrial appendage occlusion (LAAO) allows avoiding oral anticoagulation and provides at the same time an at least equally good protection from strokes and peripheral embolism. It may therefore be an attractive alternative to oral anticoagulation in the patient population undergoing transcatheter aortic valve implantation (TAVI): the concept of LAAO is based on the fact that thrombus formation in atrial fibrillation occurs in >90% in the left atrial appendage (LAA). Mechanical occlusion of the LAA reduces the stroke risk by eliminating the source of thrombus formation. In the here proposed "Randomized Comparison of Left Atrial Appendage Occlusion versus Standard Medical Therapy in Patients in Atrial Fibrillation Undergoing Transfemoral Transcatheter Aortic Valve Implantation", study we test the hypothesis, that LAAO is superior to standard medical therapy in the high-risk TAVI population. This hypothesis has not been investigated by previous studies so far.

Overall Objective(s): Overall objective: to compare the safety (and efficacy) of LAAO using the St. Jude left atrial appendage closure device with standard medical therapy in a prospective, multi-center, randomized trial in patients undergoing TAVI in routine clinical practice.

Primary Objective: To assess the safety of the device intervention with regard to stroke prevention and prevention of bleeding complications in a patients population at high risk of stroke and bleeding.

Secondary Objectives: Short-term (procedural) safety of device intervention is assessed (rate of successful deployment of a left atrial appendage occluder; rate of kidney failure). As a further secondary objective, long-term effects of device intervention on stroke and bleeding prevention as well as mortality are assessed and compared to medical therapy.

Outcome(s): Primary: Composite endpoint of ischemic and hemorrhagic neurologic events, peripheral embolism, life-threatening/disabling and major bleeding complications and cardiovascular mortality at 1 year

Secondary: All deaths (cardiac and non-cardiac) at 30 days, 1, 3, and 5 years Device success at 30 days

In-hospital acute kidney injury (AKI)

Study design: An investigator-initiated, randomized, multicenter, non-blinded, all-comers study

Measurements and Procedures: 80 patients in atrial fibrillation undergoing TAVI will be randomized in a non-blinded fashion (1:1 randomization) to LAAO (device group) or SMT at the operators' discretion (medical group; antiplatelet therapy and oral anticoagulation or oral anticoagulation alone). All patients will be followed for up to 5 years. The primary analysis will be performed at 30 days and after completion of a 1-year follow-up.

80 patients in atrial fibrillation undergoing TAVI will be randomized in a non-blinded fashion (1:1 randomization) to LAAO (device group) or standard medical therapy (SMT) at the operators' discretion (medical group; antiplatelet therapy, oral anticoagulation or oral anticoagulation alone).

Estimated duration for the main investigational plan from start of screening of first participant to last participant processed and finishing the study: 6 years

DETAILED DESCRIPTION:
Background and Rationale

Transcatheter aortic valve implantation (TAVI) is a minimally invasive treatment option for patients suffering from severe symptomatic aortic stenosis. Superiority of TAVI over medical treatment has been shown in the randomized PARTNER B trial followed by the PARTNER A trial showing non-inferiority over a more invasive open-heart surgical aortic valve replacement in high-risk patients. Over the last years, many patients have been successfully treated with TAVI worldwide.

Peri- and post-procedural morbidity differed considerably between the surgical and interventional treatment group in the PARTNER A trial: while major bleeding (19.5% vs 9.3% at 30 days) and new onset atrial fibrillation (16% vs 8.6% at 30 days) occur more often in surgically treated patients, vascular access complications (3.8 vs 17% at 30 days) and neurologic events (5.5% vs 2.4% at 30 days) are more frequently encountered in the TAVI population. The higher rate of neurologic events in the TAVI group was of particular concern, given its association with a higher mortality and the clinical impact of major neurologic events on patient's quality of life and daily functioning. Only about 40-50% of strokes occur intra-procedurally, followed by a higher hazard rate in the first week and a constant hazard thereafter. After 30 months, the surgical group experienced a numerically higher stroke rate, although not statistically significant. Measures to reduce procedural and post-procedural stroke rate were and are still looked for.

While procedural strokes can be most likely reduced by improvements in valve delivery systems (smaller delivery systems) and more operator experience, cerebral protection devices are currently tested in trials but preliminary results are rather disappointing. Risk factors for post-procedural strokes after TAVI are a previous history of stroke, more extensive peripheral vascular disease, and higher functional class.

A subgroup of patients of particular concern are patients suffering from atrial fibrillation: predictor of early (day 1-30) cerebrovascular events was new-onset atrial fibrillation (OR 2.76), whereas chronic atrial fibrillation was a predictor (OR 2.84) for the occurrence of late (>30 days) cerebrovascular events. Amat-Santos reported a higher rate of strokes/systemic embolism in patients with in hospital new onset atrial fibrillation after TAVI (13.6% vs 3.2% after 30 days). Patients diagnosed with new onset atrial fibrillation during or after the procedure in which no anticoagulation was initiated experienced an alarmingly high 30-day stroke rate of 40%.

Despite these results and the high prevalence of atrial fibrillation (AF) of about 33% in the overall TAVI population, only 30% of AF patients were on vitamin K antagonists (VKA) before, and only 70% after TAVI. While oral anticoagulation is an effective medical treatment for ischemic stroke prevention in these patients, it is often withheld from patients given their high risk of bleeding. TAVI patients typically not only suffer from much co-morbidity and are poly-medicated, but also suffer from a lot of bleeding risk factors. The bleeding risk score (HASBLED score) expresses the risk of major bleeding with a scoring system consisting of 9 individual risk factors for bleeding; a patient is at high risk for bleeding, if 3 or more factors are present. The stroke risk score (CHA2DS2-Vasc score) comprises of 9 individual risk scores for stroke in patients suffering from atrial fibrillation. Both risk scores share common risk factors, such as age, hypertension and previous stroke. It is therefore not surprising that patients at highest risk for stroke are at the same time at highest risk for major bleedings. The TAVI population forms such a high risk group with a high prevalence of the above risk factors: average patients age in the PARTNER trial was 84 years, with 11% showing severe renal impairment, about 75% had an indication for concomitant acetylsalicylic acid use and all suffered per definition from heart failure. In Stortecky's study on TAVI patients suffering AF, the average CHA2DS2-Vasc score was 4.5, with >95% of patients having a score >3.

Left atrial appendage occlusion (LAAO) allows avoiding oral anticoagulation and provides at the same time an at least equally good protection from strokes and peripheral embolism. It may therefore be an attractive alternative to oral anticoagulation in the TAVI patient population: the concept of LAAO is based on the fact that thrombus formation in atrial fibrillation occurs in >90% in the left atrial appendage (LAA). Mechanical occlusion of the LAA reduces the stroke risk by eliminating the source of thrombus formation.

Clinical studies proved this concept to be true: the PROTECT-AF study randomized >700 patients to either LAA occlusion or medical therapy (VKA). At one year, non-inferiority of LAAO was proven, with numerically less embolic events in the LAAO group. At a European conference (EuroPCR conference) 2013, Holmes (principal investigator of the PROTECT-AF trial) reported 4-year follow-up data with a significant 40% reduction of the composite of stroke/peripheral embolism/cardiovascular death and a 34% reduction of all cause mortality in the LAAO group as compared to oral anticoagulation. By reducing bleeding complications, it can be anticipated that morbidity and mortality will continue to diverge between the two groups. Comparable results from a large registry using Amplatzer devices (St. Jude Medical, St. Paul, USA) for LAAO were reported: after an average follow-up of 32 months, cardiovascular death, stroke, and peripheral embolism occurred in 7% of patients. In the latter study, oral anticoagulation was instantly stopped after LAAO in all patients.

In the here proposed "Randomized Comparison of Left Atrial Appendage Occlusion versus Standard Medical Therapy of Atrial Fibrillation in Patients Undergoing Transfemoral Transcatheter Aortic Valve Implantation", study the investigators test the hypothesis, that LAAO is superior to standard medical therapy in the high-risk TAVI population. This hypothesis has not been investigated by previous studies so far. The design is an investigator-initiated, randomized, multicenter, non-blinded, all-comers study. It is understood, that this is a pilot trial with the intention to prove safety, but which is underpowered to show superiority over medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic valve stenosis with an indication for aortic valve replacement (e.g., symptomatic patient, decreased left ventricular (LV) function)
* Suitable anatomy for transfemoral TAVI with the Portico Transcatheter Aortic Valve System (ileofemoral arterial diameter, annulus-coronary distance, annulus diameter)
* No mobile thrombus in the LA or LAA precluding LAAO
* Atrial fibrillation with a CHA2DS2-Vasc-Score >=1. No limitation regarding the nature of atrial fibrillation (paroxysmal, permanent, persistent)

Exclusion Criteria:

* Pregnancy
* Known intolerance to aspirin, heparin, contrast media or clinically manifest nickel allergy
* Inability to provide informed consent
* Mechanical heart valve or other indication for oral anticoagulation (i.e. recent pulmonary embolism)
* Contraindication for oral anticoagulation
* Currently participating in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
embolic events | 1 year
  Assessed by telephone interview
major bleeding | 1 year
  Assessed by telephone interview
cardiovascular mortality | 1 year
  Assessed by telephone interview

SECONDARY OUTCOMES:
All deaths | 30 days
  Assessed by medical chart review and telephone interview
All deaths | 1 year
  Assessed by medical chart review and telephone interview
All deaths | 3 years
  Assessed by medical chart review and telephone interview
All deaths | 5 years
  Assessed by telephone interview
Device success | 30 days
  Assessed by review of the implant procedure (fluoroscopy and echocardiography)
Acute Kidney Injury (Review of lab results: Peak value of Creatinin) | Peak value of Creatinin at 48 hour, 72 hour after Procedure
  Review of lab results in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Jakob, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jakob P, Heinz P, Gong Y, Chen M, Binder RK, Held U, Taramasso M, Paneni F, Schuetz P, Haager PK, Kasel M, Pedrazzini G, Windecker S, Moccetti M, Pilgrim T, Luscher TF, Stahli BE, Nietlispach F; TAVI-LAAO Investigators. Left Atrial Appendage Occlusion Using the Amplatzer Amulet Device in High-Risk Patients With Atrial Fibrillation Undergoing Transcatheter Aortic Valve Intervention: A Randomized Pilot Study. Struct Heart. 2025 Oct 8;9(12):100735. doi: 10.1016/j.shj.2025.100735. eCollection 2025 Dec. PMID 41321777